CLINICAL TRIAL: NCT05911854
Title: Efficacy of Multi-waved Locked System Laser Versus Cold Compression Therapy on Breast Cancer-related Lymphoedema: Randomized Controlled Trial
Brief Title: Efficacy of Multi-waved Locked System Laser Versus Cold Compression Therapy on Breast Cancer-related Lymphoedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherine Omar Abdelaziz Mohamed Elsherif, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 004539
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group (A) Multi-waved Locked System Laser group (Experimental)
  Interventions: Device: Multi-waved Locked System Laser; Other: complete decongestive therapy
- Study group (B) Cold Compression Therapy group (Experimental)
  Interventions: Device: Cold Compression therapy; Other: complete decongestive therapy
- Group (C) Control group (Active Comparator)
  Interventions: Other: complete decongestive therapy

INTERVENTIONS:
Device: Multi-waved Locked System Laser — The M6 therapy laser is a robotized multi-target device designed to treat patients suffering pathologies affecting a wide area, and to perform automatic applications.
  Other Names: M6 therapy
  Arms: Study group (A) Multi-waved Locked System Laser group
Device: Cold Compression therapy — The BioCryo Cold Compression System is a cold therapy pneumatic compression device that safely administers sequential, gradient pneumatic compression and CryoTherapy combined.
  Other Names: BioCryo Cold Compression System
  Arms: Study group (B) Cold Compression Therapy group
Other: complete decongestive therapy — Complete decongestive therapy consists of:
  * Meticulous skin care with the use of emollients
  * Using short stretch bandages or continuous wearing of a pressure garment
  * Manual lymphatic drainage therapy
  * Remedial exercises (e.g., aerobic exercise, strength training, and stretching exercises)

SUMMARY:
This study was conducted:

* To investigate the effect of MLS Laser in the management of patients with unilateral BCRL regarding lymphatic flow, volumetric measurement and HRQL assessment.
* To investigate the effect of CCT in the management of patients with unilateral BCRL regarding lymphatic flow, volumetric measurement and HRQL assessment.
* To compare the effect of MLS Laser versus CCT in the management of patients with unilateral BCRL regarding lymphatic flow, volumetric measurement and HRQL assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with unilateral BCRL.
* Age of patients above 18 years old
* Patient history of modified radical mastectomy, chemotherapy and/or radiotherapy.
* Patients undertaken have history or current hormonal treatment.
* Patients with moderate lymphoedema (20-40% increase in extremity volume)

Exclusion Criteria:

* Patients who have severe co-morbid diseases.
* Presence of other cancers, cancer recurrence, lymphatic malformation, or vascular disease
* Patients who are having current chemotherapy and/or radiotherapy.
* Patients who have bilateral lymphedema, current metastases, elephantiasis, infection, lymphangiosis carcinomatosa, cellulitis, venous thrombosis, or congestive heart failure
* Patients with musculoskeletal disorders affecting upper extremity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change in lymphatic flow using lymphoscintigraphy pre and post treatment | Baseline
  Interpretation of the results of the lymphoscintigraphy and using the contralateral limb as a healthy control with normal lymphatic function can differentiate the lymphatic flow abnormalities into 7 stages
The change of Volumetric measurement of the arm pre and post treatment | Baseline
  Precise arm volume measurement is capital in the follow-up of breast cancer patients, as an early detection of BCRL can reduce the incidence of irreversible stages

SECONDARY OUTCOMES:
The change of Lymphedema Life Impact Scale scores pre and post treatment | Baseline
  The Lymphedema Life Impact Scale is a lymphedema-specific tool which measures physical (pain, heaviness, tightness, strength…), psychosocial (body image, socializing, intimate relations…) and functional (duties at home, duties at work, recreational activities…) impact upon the patients' lives, the maximum score is 68 while the minimum score is 0, where a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H El-Gendy, professor, Study Chair — Cairo University
Locations (1):
- Kasr El-Einy Center of Radiation Oncology and Nuclear Medicine, Faculty of Medicine, Cairo University, Cairo, Egypt